CLINICAL TRIAL: NCT02222623
Title: Insulin Glargine vs NPH as Basal Insulin on Glycemic Values in Hospitalized Patients: The Inova Diabetes Study
Brief Title: The Inova Type 2 Diabetes Mellitus Study
Acronym: InovaDM2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1623
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes, Type 2
Keywords: insulin; basal; diabetes; hospital; glucose; hypoglycemia; glargine; NPH; neutral protamine hagedorn
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus; Hypoglycemia | interventions — Insulin Glargine; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- glargine insulin (Active Comparator): Basal glargine given once daily in the morning before breakfast plus standard hospital corrective doses of insulin aspart before meals and at bedtime.
  Interventions: Drug: Glargine
- NPH insulin (Active Comparator): Basal NPH given twice daily before breakfast and at bedtime plus standard hospital corrective doses of insulin aspart before meals and at bedtime.
  Interventions: Drug: NPH

INTERVENTIONS:
Drug: Glargine — Glargine given as 100% total daily dose with breakfast. The initial dose will be calculated using the patient's weight or using their basal insulin doses prior to hospitalization.
  Other Names: Lantus
  Arms: glargine insulin
Drug: NPH — NPH 2/3 of the total daily dose given with breakfast, 1/3 of the total daily dose given at bedtime. The initial dose is calculated using the patient's weight or using the basal insulin dose prior to hospitalization.
  Other Names: Novolin N; Humulin N
  Arms: NPH insulin

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the two different basal insulins commonly used for basal blood sugar control in the treatment of type 2 diabetes mellitus in patients who are hospitalized and require low doses of insulin: neutral protamine Hagedorn (NPH) insulin and glargine (Lantus®) insulin. Previous research has shown that both NPH insulin and glargine (Lantus®) insulin is safe and effective for the control of blood sugar in a type 2 diabetic patient. This research is being done because the costs of medications for diabetic patients are very expensive. Our goal with this research is to show that a less expensive insulin (NPH) is as safe and effective as a more expensive insulin [glargine (Lantus®)] in patients with type 2 diabetes mellitus who are in the hospital.

DETAILED DESCRIPTION:
This is a randomized, open label trial comparing effectiveness of insulin glargine and insulin NPH in a basal plus correctional regimen. Patients will be randomized to either an intervention (NPH) or a control group (glargine) upon admission. The following data will be collected: age, sex, weight, preadmission diabetes medications, admission diagnosis, HbA1C, blood glucose (BG), chemistry, hematology, urine analysis, pregnancy test, duration of hospitalization, insulin dose, and discharge status. Data will be recorded and maintained confidentially.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ages18-75 admitted to a general medicine or surgical Department of Medicine hospitalist services.
2. A known history of T2DM, receiving either diet alone, low dose insulin (≤0.4 units/kg/day), OADs, GLP1 analogs, or in any combination of OADs, GLP1 analogs and low dose insulin (≤0.4 units/kg/day).
3. Subjects must have a BG >140 mg/dL and ≤240 mg/dL before randomization without laboratory evidence of diabetic ketoacidosis or hyperglycemic hyperosmolar nonketotic syndrome (bicarbonate <18 mEq/L, pH <7.30, or positive serum or urinary ketones, BG >240 mg/dL).

Exclusion Criteria:

1. Patients with a diagnosis of type 1 diabetes mellitus.
2. Patients using nutritional bolus insulin at home.
3. Patients with increased blood glucose concentration, but without a known history of diabetes.
4. Patients with a history of diabetic ketoacidosis, hyperglycemic hyperosmolar nonketotic syndrome, or ketonuria.
5. Patients admitted to or expected to require admission to any intensive care unit (ICU) or intermediate care unit (IMC).
6. Patients who are receiving or are anticipated to receive enteral or parenteral nutrition.
7. Patients admitted for cardiac surgery.
8. Patients receiving continuous insulin infusion.
9. Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, or impaired renal function (creatinine ≥ 3.5 mg/dL).
10. Persons with decisional incapacity (mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study).
11. Female subjects who are pregnant or immediately (same hospitalization) post partum at time of enrollment into the study.
12. Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mean daily blood glucose | 5 days

SECONDARY OUTCOMES:
Percent of total BG readings within target BG 70-180 mg/dL before meals. | 5 days
Number (Percent) of episodes and total BG readings of hypoglycemic events (BG < 70 mg/dL) | 5 days
Number (Percent) of total BG readings of severe hyperglycemia (BG > 300 mg/dL) after the first day of treatment. | 5 days
Hospital mortality | 5 days

OTHER OUTCOMES:
Mean total daily dose of insulin | 5 days
Length of hospital stay | within first 30 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Clement, MD, Principal Investigator — Inova Fairfax Hospital
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States